CLINICAL TRIAL: NCT00782691
Title: Validation of FDG-PET Segmentation Tools for Tumor Delineation by Correlation of CT- and FDG-PET Volume Measurements With Histopathology of Nodal Metastases of Head and Neck Carcinomas.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: D.A.X. Schinagl, Radboud University Nijmegen Medical Centre
Other Study IDs: 2008/060
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Head and Neck Cancer
Keywords: FDG-PET segmentation tools; Head-and-neck cancer; Histological validation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Head-and-neck cancer patients will undergo a therapeutic lymph node dissection of the cervical nodes. This treatment is given whether the patient is enrolled in the study or not. Histological specimens of cancer patients are always stored for possible future refference in the routine clinical practice.

GROUPS / COHORTS (1):
- Head-and-neck cancer patients.: Head-and-neck cancer patients eligible for therapeutic lymph node dissection of cervical nodes.
  Interventions: Other: CT-FDG/PET scan of the head-and-neck region

INTERVENTIONS:
Other: CT-FDG/PET scan of the head-and-neck region — CT-FDG/PET scan of the head-and-neck region

SUMMARY:
Various methods of FDG-PET signal segmentation will be validated by correlation of histopathologically measured tumor dimensions in lymph node dissection specimens of head-and-neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with N+ squamous cell carcinoma of the head and neck, planned for neck dissection.
* Age >18 years.

Exclusion Criteria:

* Pregnancy.
* Women breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head-and-neck cancer patients eligible for therapeutic lymph node dissection of cervical nodes.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
How accurate are the various FDG-PET segmentation tools? | Measurements are performed in conjunction with the clinical pathologist directly postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands